CLINICAL TRIAL: NCT02956499
Title: A First-in-Human, Randomized, Dose-Escalation, Double-Blind, Placebo-Controlled Study to Assess Safety, Tolerability and Pharmacokinetics of APX001 Administered by Intravenous Infusion to Healthy Subjects
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics of APX001 Administered by Intravenous Infusion to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: APX001-101; C4791001 (Other: Alias Study Number)
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1 (Experimental): single intravenous dose
  Interventions: Drug: APX001 single dose 1; Drug: Matching Placebo
- Cohort 2 (Experimental): single intravenous dose
  Interventions: Drug: APX001 single dose 2; Drug: Matching Placebo
- Cohort 3 (Experimental): single intravenous dose
  Interventions: Drug: APX001 single dose 3; Drug: Matching Placebo
- Cohort 4 (Experimental): single intravenous dose
  Interventions: Drug: APX001 single dose 4; Drug: Matching Placebo
- Cohort 5 (Experimental): single intravenous dose
  Interventions: Drug: APX001 single dose 5; Drug: Matching Placebo
- Cohort 6 (Experimental): single intravenous dose
  Interventions: Drug: APX001 single dose 6; Drug: Matching Placebo
- Cohort 7 (Experimental): multiple intravenous doses
  Interventions: Drug: APX001 multiple dose 1; Drug: Matching Placebo
- Cohort 8 (Experimental): multiple intravenous doses
  Interventions: Drug: APX001 multiple dose 2; Drug: Matching Placebo
- Cohort 9 (Experimental): multiple intravenous doses
  Interventions: Drug: APX001 multiple dose 3; Drug: Matching Placebo
- Cohort 10 (Experimental): multiple intravenous doses
  Interventions: Drug: APX001 multiple dose 4; Drug: Matching Placebo

INTERVENTIONS:
Drug: APX001 single dose 1
  Arms: Cohort 1
Drug: APX001 single dose 2
  Arms: Cohort 2
Drug: APX001 single dose 3
  Arms: Cohort 3
Drug: APX001 single dose 4
  Arms: Cohort 4
Drug: APX001 single dose 5
  Arms: Cohort 5
Drug: APX001 single dose 6
  Arms: Cohort 6
Drug: APX001 multiple dose 1
  Arms: Cohort 7
Drug: APX001 multiple dose 2
  Arms: Cohort 8
Drug: APX001 multiple dose 3
  Arms: Cohort 9
Drug: APX001 multiple dose 4
  Arms: Cohort 10
Drug: Matching Placebo

SUMMARY:
First In Human (FIH), randomized, double-blind, placebo-controlled single ascending dose (SAD) and multiple ascending dose (MAD) escalation study of approximately 80 subjects. The SAD portion of the study will enroll six cohorts of eight healthy subjects per cohort, for a total of approximately 48 healthy subjects. The MAD portion of the study will enroll four cohorts of eight healthy subjects per cohort, for a total of approximately 32 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must agree to avoid pregnancy during the study and to use contraception at least 2 weeks before the start of the study until 3 months after the last dose of study drug.
* Males with partner(s) of childbearing potential must agree to use appropriate barrier contraception from the screening period until 3 months after the last dose of study drug.
* Screening hematology, clinical chemistry, coagulation and urinalysis consistent with overall good health.
* No significantly abnormal findings on physical examination, ECG and vital signs.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Any uncontrolled or active major systemic disease including, but not limited to: cardiovascular, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential.
* History or presence of malignancy within the past year. Subjects who have been successfully treated with no recurrence of basal cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
* Use of prescription medication within 14 days prior to the first dose of study drug and throughout the study.
* Use of non-prescription or over-the-counter medications within 7 days prior to the first dose of study drug and throughout the study.
* Positive results on any of the following Screening laboratory tests: serum pregnancy test, urine alcohol test, urine drugs of abuse, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of APX001 as measured by adverse events (AEs), physical examinations (PE), vital signs (VS), laboratory safety tests, urinalysis and 12-lead electrocardiograms (ECG). | 21 days

SECONDARY OUTCOMES:
Pharmacokinetics of single and multiple doses of APX001 as measured by maximum observed concentration (Cmax). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by area under the curve (AUC). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by terminal phase half-life (t1/2). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by volume of distribution (Vd). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by elimination rate constant (Kel). | 21 days
Pharmacokinetics of single and multiple dose of APX001 as measured by accumulation ratio. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodges MR, Ople E, Wedel P, Shaw KJ, Jakate A, Kramer WG, Marle SV, van Hoogdalem EJ, Tawadrous M. Safety and Pharmacokinetics of Intravenous and Oral Fosmanogepix, a First-in-Class Antifungal Agent, in Healthy Volunteers. Antimicrob Agents Chemother. 2023 Apr 18;67(4):e0162322. doi: 10.1128/aac.01623-22. Epub 2023 Mar 29. PMID 36988461